CLINICAL TRIAL: NCT06896591
Title: Effets D'un Bloc Glutéal Postérieur Profond Associé À Un PENG Bloc Dans La Prothèse Totale De Hanche
Brief Title: Deep Posterior Post Gluteal Compartment Block in Total Hip Arthroplasty: Feasability and Safety
Acronym: ANATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quincy Anesthésie (Network)
Responsible Party: Principal Investigator, Yoann ELMALEH, Medical Doctor, Anesthesiology and Pain Medicine, Principal Investigator, Quincy Anesthésie
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COS-RGDS-2024-06-039-P-ELMALEH
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Total Hip Arthroplasty
Keywords: total hip arthroplasty; peng block; Hip; Anatomy; Sciatic nerve block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DPPG compartment block (Experimental): Deep posterior post gluteal compartment block with different volume of product 5,10 and 15 ml (local anesthetics such as naropeine 0.35%) to compare the efficiency of the block without sciatic nerve block effect
  Interventions: Procedure: Deep posterior post gluteal nerve block

INTERVENTIONS:
Procedure: Deep posterior post gluteal nerve block — One injection with ultrasound guidance injection of 5, 10 or 15 mL of naropeine 0.35 % Procedure : injection below the piriformis muscle in front of the head of the femur.

SUMMARY:
This study aims to evaluate the effectiveness of a posterior hip capsule block performed in addition to a PENG (Pericapsular Nerve Group) block for patients undergoing hip arthroplasty. The primary objective is to assess whether this combined approach provides enhanced perioperative analgesia compared to the standard analgesic protocol or the PENG block alone. Secondary outcomes will focus on opioid consumption, functional recovery, and any potential complications. By targeting both the anterior and posterior innervation pathways around the hip joint, this combined technique could improve patient comfort, decrease opioid requirements, and potentially expedite rehabilitation after hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

All adults with total hip arthroplasty

-

Exclusion Criteria:

* Contraindication to regional anesthesia
* allergy
* refusal of the injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sciatic nerve block | From enrollment to the end of treatment at 1 month
  number of patients with postoperative sciatic motor or sensitory nerve block collected by clinical examination (test with hot and cold in the sciatic territory and motricity of the feet)

SECONDARY OUTCOMES:
Pain postoperative | From enrollment to the end of treatment at 1 MONTH
  Visual analogic pain (VAS) AT 6 hours 0 : no pain 10: maximum pain
pain 2 | From enrollment to the end of treatment at 1 MONTH
  Visual analogic pain (VAS) AT 12 hours 0 : no pain 10: maximum pain
oPIOID Consumption | From enrollment to the end of treatment at 7 months
  Opioid consumption per and postoperative until 48 hours
RAAC | From enrollment to the end of treatment at 1 MONTH
  QOR15 scale at H24 and H48 questionnaire with 15 questions from 0 to 10 (https://pqip.org.uk/FilesUploaded/Myles%20QoR-15.pdf)
Surgical complication | From enrollment to the end of treatment at 1 MONTH
  Surgical postoperative complication or fall

CONTACTS AND LOCATIONS:
Overall Officials: yoann ELMALEH, M.D, Principal Investigator — Hopital Privé Claude Galien

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pun M, Ng T, Vermeylen K, Tran J. Innervation of the hip joint: implications for regional anaesthesia and image-guided interventional pain procedures. BJA Educ. 2024 Jun;24(6):191-202. doi: 10.1016/j.bjae.2024.02.005. Epub 2024 Apr 8. No abstract available. PMID 38764441